CLINICAL TRIAL: NCT05941065
Title: Open-label, Prospective Study of Skin Balancing Gel Cream Safety and Influence of Skin Microbiome on Acne Prone Skin
Brief Title: Study of Skin Balancing Gel Cream Safety and Influence of Skin Microbiome on Acne Prone Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Burt's Bees Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BB_SKIN_BALANCE
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Skin Microboime; Acne
Keywords: Skin; Microbiome
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balancing gel cream (Experimental): Product will be used twice daily in the morning and in the evening for 6 weeks. 1-2 pumps (dime size) of product will be applied on the face.
  In addition to the study product, a Cetaphil cleanser will be used as well. Cleanser will be applied twice daily in the morning and in the evening for 6 weeks. Cleanser will be used on wet face and gently pat dry.
  Interventions: Other: Balancing gel cream

INTERVENTIONS:
Other: Balancing gel cream — Skin balancing gel cream will be applied onto clean skin morning and night

SUMMARY:
The purpose of this study is to assess the safety of the skin balancing gel cream and examine the effects it has on the skin microbiome of individuals with non-cystic acne prone skin.

DETAILED DESCRIPTION:
Acne, a chronic inflammatory condition, is estimated to affect greater than 85% of the population at some point. It is considered a common skin condition characterized by pimples and occurs when follicles are clogged leading to the formation of acne lesions. In this study, we want to evaluate the impact the skin balancing gel cream has on the skin microbiome on individuals who have mild to moderate non-cystic acne. We will be assessing the changes it has on specific microbiota (Cutibacterium acnes for example) and whether it is tolerated well on acne prone skin.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between the ages of 18 years of age until 35 years of age
* Males must be willing to shave facial hair
* The presence of mild to moderate non-cystic acne based on investigator global assessment

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners.
* Adults unable to consent.
* The presence of severe acne or cysts as noted by the investigator.
* Those who are unwilling to discontinue topical antibiotics, topical salicylic acid containing products and topical benzoyl peroxide containing products for two weeks to meet the washout criteria prior to enrolling.
* Those who are unwilling to discontinue all facial topical products except the cleanser and the product provided in the study.
* Individuals who have been on an oral antibiotic for acne within the previous 1 month.
* Individuals who have changed any of their hormonal based contraception within 3. months prior to joining the study.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
C. acnes relative abundance | 6 weeks
  Shift in the C. acnes relative abundance based on skin microbiome swab collection and sequencing

SECONDARY OUTCOMES:
Functional gene based predictive analysis of skin inflammation related genes | 6 weeks
  Functional gene analysis for skin inflammation related genes from whole genome sequencing of facial skin microbiome
Sebum excretion rate | 6 weeks
  Measure of skin sebum via sebumeter
Tolerability Assessment Questionnaire | 6 weeks
  A 6 question survey based on the self-assessment about the tolerability of the topical skin product such as itching, burning, and stinging. The scale ranges from 0-3 with 0 being the best outcome possible and with 3 being the worst.
  "0" as none, "1" as mild, "2" as moderate, or "3" as severe.
Total lesion count | 6 weeks
  Safety endpoint to count inflammatory and non-inflammatory lesions to ensure that there is not a flare in the acne

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD MS AP, Principal Investigator — Integrative Skin Science and Research
Locations (1):
- Integrative Skin and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No